CLINICAL TRIAL: NCT04677491
Title: Effects of Ospemifene on Brain Activation Patterns in Women With Sexual Interest-arousal Disorders
Acronym: EROS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Camil Castelo-Branco, Principal Investigator, Clinical Professor, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2020-001514-38
Record Dates: First submitted 2020-11-23; First posted 2020-12-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2022-02

CONDITIONS: Vulvovaginal Signs and Symptoms; Genitourinary Syndrome of Menopause; Sexual; Disorder, Arousal, Female
Keywords: Sexual Disorder; Genitourinary Syndrome of Menopause
MeSH Terms: conditions — Coitus; Sexual Dysfunction, Physiological | interventions — Ospemifene

STUDY DESIGN:
Intervention Model Description: Pilot study, randomised prospective study, triple blind, placebo controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VVA-FSIAD ospemifene group (Active Comparator): Women treated with ospemifene 60 mg/day
  Interventions: Drug: Ospemifene 60 mg; Behavioral: fMRI experiments
- VVA-FSIAD placebo group (Placebo Comparator): Women treated with placebo
  Interventions: Behavioral: fMRI experiments

INTERVENTIONS:
Drug: Ospemifene 60 mg — Ospemifene vs placebo
  Other Names: Senshio
  Arms: VVA-FSIAD ospemifene group
Behavioral: fMRI experiments — Participants will see sexually explicit video clips that alternate with non-sexual clips and neutral color projection and b) smell alternate pheromones with clear air and pine aroma.

SUMMARY:
Ospemifene is the first oral and non-hormonal treatment for moderate or severe vulvo-vaginal atrophy (VVA) in postmenopausal women who are not candidates to treatment with local oestrogens. Its effects are mediated though the regeneration of the proportion of superficial and intermediate cells of the vagina, improving menopausal symptomatology such as dryness and dyspareunia.

Only two studies to date have directly compared brain activation patterns in women with normal sexual function with women complaining with hypoactive sexual desire disorder. Arnow et al. demonstrated that women with normal sexual function showed brain activations in multiple regions different from women with FSIAD. When comparing the two groups, women with normal sexual function showed greater activation of the bilateral entorhinal cortex while women with FSIAD exhibited greater activation of the medial frontal gyrus, right inferior frontal gyrus, and bilateral putamen. The medial frontal gyrus activation has been associated with self-monitoring; thus, it is possible that women with FSIAD allocate more attention to monitoring their response, which may be inhibitory to sexual functioning. The other study was done by Woodard and colleges showing that women with normal sexual function showed significantly differences on cerebral activation in comparison with women with FSIAD.

These differences observed in women with FSIAD could suggest that they may have alterations in activation of limbic and cortical structures responsible for acquiring, encoding, and retrieving memory, the processing and memory of emotional reactions, and areas responsible for heightened attention to one's own physical state.

For this reason the authors believe that it is essential to determine if the effect of ospemifene on the improvement on sexual function is due to the improvement on the vagina tract or due to its effect on brain function.

DETAILED DESCRIPTION:
To evaluate changes from baseline in brain activation patterns, by using functional magnetic resonance imaging (fMRI) techniques and sexual stimuli, in postmenopausal women with moderate to severe vulvovaginal atrophy and FSIAD after 3 months treatment with ospemifene 60mg/day compared to those treated with placebo. fMRI technique allows the study of brain activation by detecting brain blood flow and oxygen level dependent changes induced by neuronal activation.

The brain activation patterns will be defined by the number of voxels that significantly changed their signal intensity during the stimuli presentation compared to the neutral stimuli. Brain connectivity will be evaluated by using the activation map and the atlas of neuroanatomic regions and comparing the number of voxels, its level of significance and the different regions activated.

Brain activation patterns changes (with fMRI) after sexual stimuli (visual or olfactive), in postmenopausal women with moderate to severe VVA and FSIAD after 3 months treatment with ospemifene 60mg/day compared to those treated with placebo.

During the fMRI session, the activation of each brain circuits/pattern is measured by the blood-oxygen level dependent (BOLD) signal and with the Statistical Parametric Mapping method regularly used in fMRI studies to visualize brain activation.

For the longitudinal study, a paired t-test will be used within each group to detect changes in activation over time. The statistical threshold criterion to compare the different activation maps between both groups is p < 0.001 uncorrected with a minimum extent of 10 voxels. Only clusters that survive a p < 0.05 FWE (family wise error) correction for multiple comparisons will be considered statistically significant The region of interests who were mainly observed are: medial occipital gyrus, anterior cingulate cortex, bilateral thalamus, caudate nucleus, left pale globe, cerebellum, left inferior parietal lobe, postcentral gyrus, praecuneus, right medial frontal gyrus and left praecuneus.

A total of 20 consecutive postmenopausal women with moderate to severe VVA and FSIAD with symptomatology will be recruited to participate in the study, 10 of which will be randomised to the ospemifene group (VVA-FSIAD ospemifene group) and 10 will be randomised to the placebo group (VVA-FSIAD placebo group). Additionally, a total of 5 consecutive postmenopausal women with moderate to severe VVA not treated with ospemifene neither with any other VVA treatment and without FSIAD will also be recruited (VVA not treated patients without FSIAD).

ELIGIBILITY:
Inclusion criteria:

* Women 40 year old or older who have been diagnosed with menopause (either chemical, surgical or natural menopause)
* No menstruation for at least a year.
* Moderate or severe VVA diagnosis (defined by the presence of ≤ 5% of superficial cells and vaginal pH > 5).
* For homogenisation of brain patterns, women had to be right-handed.
* Women should be strictly heterosexual, in a stable relationship of at least 1 year duration (with expectations of remaining with the same relationship), and have had experience viewing sexually explicit images
* For the FSIAD groups, women will be included if they are diagnosed with FSIAD, defined according to the criteria of DSM-V and confirmed by a structured clinical interview and by means of the scores of the SFQ and the FSDS-R (with a score of ≤20 for FSFI and ≥15 for the FSDS-R, respectively). These criteria will be an exclusion criterion for women without FSIAD.
* Informed written consent of the patient.

Exclusion criteria

* Women with known history of mental illness, history of drug or alcohol abuse.
* Women with VVA treatment (oestrogens or ospemifene) at any time during the last 6 months, and/or laser treatment at any time during the last year.
* Use of medication or herbal preparations at any time during the last 3 months for the purpose of improving sexual performance.
* Women who have received any medication previous to the study inclusion, that may alter or interfere with brain activation patterns (psychoactive drugs).
* Women with history of sexual offenses.
* Women with abnormal vision that would impair the visualisation of the images and the olfactory stimuli.
* Women with claustrophobia or implants that would preclude fMRI procedures.
* Women with diagnosis of depression assessed by PHQ self-administered questionnaire.
* Patients who had undergone vaginal surgery in the last 12 months.
* Women who did not sign the written informed consent.
* Hypersensitivity to the active substance or to any of the excipients included in Senshio.
* Past or active history of venous thromboembolic events (VTE), including deep vein thrombosis, pulmonary embolism and retinal vein thrombosis.
* Unexplained vaginal bleeding.
* Patients with suspected breast cancer or who are receiving active treatment (including adjuvant treatment) for breast cancer.
* Suspicion of neoplasia or active neoplasia dependent on sex hormones (eg endometrial cancer).
* Patients with signs or symptoms of endometrial hyperplasia; In this group of patients, safety has not been studied.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
a Activation of each brain circuits | 3 months
  Is measured by the blood-oxygen level dependent (BOLD)

SECONDARY OUTCOMES:
Vaginal pH | 3 months
  vaginal pH measured by ph roll from 1 to 14
Vaginal maturation index | 3 months
  vaginal maturation index meadured by vaginal citology on percentage from 0 to 100 divided in superficial, intermediate and basal cells
Vaginal health index | 3 months
  To describe if there is a correlation between changes in the visual examination of the vagina. using the vaginal health index: from 5 to 25 (min-max).
Female Sexual Function Index | 3 months
  Questionaire from 18 to 90 (min-max).
DSM V evaluation | 3 months
  DSM Criteria
Quality of Life Scale | 3 months
  Questionaire PHQ9 (Patient health questionaire 9) from 0 to 27 (min-max)
Female Sexual Distress Scale | 3 months
  Questionaire FSFI (Female Sexual Function Index) from 18 to 90 (min-max).
Social Functioning Questionnaire | 3 months
  Questionaire SF12 (Physical and Mental Health Composite Scores) from 0 to 12 (min-max)
Patient Health Questionnaire-9 | 3 months
  Questionaire from 0 to 9

CONTACTS AND LOCATIONS:
Overall Officials: Camil Castelo-Branco, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No